CLINICAL TRIAL: NCT03909841
Title: Neuropathic Pain in Elderly People With Diabetes: Impact on Quality of Life and Cognition
Status: Completed | Type: Observational
Sponsor: Queen Elizabeth Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Woo Cheuk Wai, Physiotherapist, Queen Elizabeth Hospital, Hong Kong
Other Study IDs: KC/KE-17-0070/ER-1
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus; Diabetic Peripheral Neuropathy; Cognitive Impairment; Quality of Life; Diabetic Peripheral Neuropathic Pain
MeSH Terms: conditions — Diabetes Mellitus; Cognitive Dysfunction | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DM: DM without DPN (Diabetic Peripheral Neuropathy)
  Interventions: Behavioral: Cambridge Neuropsychological Test Automated Battery (CANTAB); Other: Chinese (Hong Kong) 12-item Short-Form Health Survey (version 2)
- DPN: DM with DPN (Diabetic Peripheral Neuropathy)
  Interventions: Behavioral: Cambridge Neuropsychological Test Automated Battery (CANTAB); Other: Chinese (Hong Kong) 12-item Short-Form Health Survey (version 2)
- DPN-P: DM with DPN-P (Diabetic Peripheral Neuropathic Pain)
  Interventions: Behavioral: Cambridge Neuropsychological Test Automated Battery (CANTAB); Other: Chinese (Hong Kong) 12-item Short-Form Health Survey (version 2)

INTERVENTIONS:
Behavioral: Cambridge Neuropsychological Test Automated Battery (CANTAB) — Cognition using Cambridge Neuropsychological Test Automated Battery (CANTAB)
Other: Chinese (Hong Kong) 12-item Short-Form Health Survey (version 2) — Quality of Life using Chinese (Hong Kong) 12-item Short-Form Health Survey (version 2)

SUMMARY:
This study was set out 1) Evaluate the impact of Diabetic Peripheral Neuropathy (DPN) and DPN-P (Diabetic Peripheral Neuropathic Pain) on the overall Quality of Life (QoL) in elderly with Diabetic Mellitus (DM) and 2) Evaluate the association between cognition impairments and DM in the elderly, and the contributions of DPN and/or DPN-P

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 or above
* Diagnosis of diabetes mellitus (Type 1 or Type 2)

Exclusion Criteria:

* major psychiatric conditions
* recent cardiovascular events within the last six months
* blindness radiculopathy
* spinal cord injury, multiple sclerosis
* carpal tunnel syndrome
* trigeminal neuralgia
* Subjects who were incompetent in giving written consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with Diabetes Mellitus attending the diabetes clinic and / or pain clinic
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Cognition | Day 1
  Identifying cognitive affected domains by using Cambridge Neuropsychological Test Automated Battery (CANTAB) (Reaction Time : RTI, Spatial Working Memory : SWM and Executive Function : OTS)

SECONDARY OUTCOMES:
Quality of Life: The Chinese (Hong Kong) 12-item Short-Form Health Survey version 2 | Day 1
  Identifying Quality of Life affected domains by using The Chinese (Hong Kong) 12-item Short-Form Health Survey version 2

CONTACTS AND LOCATIONS:
Overall Officials: Research Ethics Committee (Kowloon Central/ Kowloon East), Study Chair — Research Ethics Committee (Kowloon Central/ Kowloon East)
Locations (1):
- Queen Elizabeth Hospital, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No